CLINICAL TRIAL: NCT01065012
Title: Open-Label Phase 3 Study to Evaluate the Long-Term Safety and Efficacy of Udenafil Tablets in Male Subjects With Erectile Dysfunction
Brief Title: Treatment of Erectile Dysfunction - Long Term Safety and Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-01409
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Udenafil 50 mg (Experimental): 50 mg Udenafil
  Interventions: Drug: Udenafil 50 mg; Drug: Placebo Matching 100 mg Udenafil; Drug: Placebo Matching 150 mg Udenafil
- Udenafil 100 mg (Experimental): 100 mg Udenafil
  Interventions: Drug: Udenafil 100 mg; Drug: Placebo Matching 50 mg Udenafil; Drug: Placebo Matching 150 mg Udenafil
- Udenafil 150 mg (Experimental): 150 mg Udenafil
  Interventions: Drug: Udenafil 150 mg; Drug: Placebo Matching 50 mg Udenafil; Drug: Placebo Matching 100 mg Udenafil
- Placebo (Placebo Comparator): Placebo Tablets matching Udenafil tablets
  Interventions: Drug: Placebo Matching 50 mg Udenafil; Drug: Placebo Matching 100 mg Udenafil; Drug: Placebo Matching 150 mg Udenafil

INTERVENTIONS:
Drug: Udenafil 50 mg — Tablets via oral administration before an attempt at sexual intercourse. All subjects started at 100 mg and titrated up to 150 mg or down to 50 mg per Investigator and subject.
  Other Names: WC3043
  Arms: Udenafil 50 mg
Drug: Udenafil 100 mg — Tablets via oral administration before an attempt at sexual intercourse. All subjects started at 100 mg and titrated up to 150 mg or down to 50 mg per Investigator and subject.
  Other Names: WC3043
  Arms: Udenafil 100 mg
Drug: Udenafil 150 mg — Tablets via oral administration before an attempt at sexual intercourse. All subjects started at 100 mg and titrated up to 150 mg or down to 50 mg per Investigator and subject.
  Other Names: WC3043
  Arms: Udenafil 150 mg
Drug: Placebo Matching 50 mg Udenafil — Tablets via oral administration before an attempt at sexual intercourse. All subjects started at 100 mg and titrated up to 150 mg or down to 50 mg per Investigator and subject.
  Other Names: Placebo 50 mg
  Arms: Placebo; Udenafil 100 mg; Udenafil 150 mg
Drug: Placebo Matching 100 mg Udenafil — Tablets via oral administration before an attempt at sexual intercourse. All subjects started at 100 mg and titrated up to 150 mg or down to 50 mg per Investigator and subject.
  Other Names: Placebo 100 mg
  Arms: Placebo; Udenafil 150 mg; Udenafil 50 mg
Drug: Placebo Matching 150 mg Udenafil — Tablets via oral administration before an attempt at sexual intercourse. All subjects started at 100 mg and titrated up to 150 mg or down to 50 mg per Investigator and subject.
  Other Names: Placebo 150 mg
  Arms: Placebo; Udenafil 100 mg; Udenafil 50 mg

SUMMARY:
Open-Label Phase 3 study to evaluate the long-term safety and efficacy of udenafil, an orally administered selective inhibitor of PDE-5 for the treatment of subjects with erectile dysfunction (ED).

DETAILED DESCRIPTION:
Patients completing the double-blind phase will be entered into Study 01409 at the intermediate dose. Up and down dose adjustments will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed Study PR-01209 or PR-01309
* Continues in a stable monogamous relationship with a consenting female partner who is at least 19 years of age.
* Partner is not pregnant or lactating

Exclusion Criteria:

* Symptomatic coronary artery disease, myocardial infarction or cardiac surgical procedure.
* Cardiac arrhythmias requiring antiarrhythmic treatment
* Symptomatic congestive heart failure
* Taking nitrate medication in any form
* Uncontrolled diabetes (HbA1c ≥ 13%)
* Hypersensitivity to phosphodiesterase type 5 (PDE-5) inhibitors

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) score | Assessment will be made after each use of the study drug over a 36 week use period.

SECONDARY OUTCOMES:
Changes in the satisfaction of intercourse, orgasmic function, sexual desire and overall satisfaction | Assessment will be made after each use of the study drug over a 36 week use period.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (69):
- United States (69):
  - Warner Chilcott Investigational Site, Birmingham, Alabama
  - Warner Chilcott Investigational Site, Homewood, Alabama
  - Warner Chilcott Investigational Site, Huntsville, Alabama
  - Warner Chilcott Investigational Site, Mesa, Arizona
  - Warner Chilcott Investigational Site, Phoenix, Arizona
  - Warner Chilcott Investigational Site, Tempe, Arizona
  - Warner Chilcott Investigational Site, Tucson, Arizona
  - Warner Chilcott Investigational Site, Chino, California
  - Warner Chilcott Investigational Site, Laguna Hills, California
  - Warner Chilcott Investigational Site, Newport Beach, California
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Tarzana, California
  - Warner Chilcott Investigative Site, Torrance, California
  - Warner Chilcott Investigational Site, Denver, Colorado
  - Warner Chilcott Investigational Site, Englewood, Colorado
  - Warner Chilcott Investigational Site, Middlebury, Connecticut
  - Warner Chilcott Investigational Site, Milford, Connecticut
  - Warner Chilcott Investigative Site, New Britain, Connecticut
  - Warner Chilcott Investigational Site, Waterbury, Connecticut
  - Warner Chilcott Investigational Site, Aventura, Florida
  - Warner Chilcott Investigational Site, Clearwater, Florida
  - Warner Chilcott Investigational Site, Daytona Beach, Florida
  - Warner Chilcott Investigational Site, DeLand, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Ocala, Florida
  - Warner Chilcott Investigational Site, Tampa, Florida
  - Warner Chilcott Investigational Site, Columbus, Georgia
  - Warner Chilcott Investigational Site, Dawsonville, Georgia
  - Warner Chilcott Investigational Site, Sandy Springs, Georgia
  - Warner Chilcott Investigational Site, Melrose Park, Illinois
  - Warner Chilcott Investigational Site, Fort Wayne, Indiana
  - Warner Chilcott Investigational Site, Greenwood, Indiana
  - Warner Chilcott Investigational Site, Jeffersonville, Indiana
  - Warner Chilcott Investigational Site, West Des Moines, Iowa
  - Warner Chilcott Investigational Site, Elkridge, Maryland
  - Warner Chilcott Investigational Site, Omaha, Nebraska
  - Warner Chilcott Investigational Site, Las Vegas, Nevada
  - Warner Chilcott Investigational Site, Lawrenceville, New Jersey
  - Warner Chilcott Investigational Site, Bay Shore, New York
  - Warner Chilcott Investigational Site, Garden City, New York
  - Warner Chilcott Investigational Site, Kingston, New York
  - Warner Chilcott Investigational Site, New York, New York
  - Warner Chilcott Investigational Site, Poughkeepsie, New York
  - Warner Chilcott Investigational Site, Rochester, New York
  - Warner Chilcott Investigational Site, Williamsville, New York
  - Warner Chilcott Investigational Site, Cary, North Carolina
  - Warner Chilcott Investigational Site, Concord, North Carolina
  - Warner Chilcott Investigational Site, Harrisburg, North Carolina
  - Warner Chilcott Investigational Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Site, Salisbury, North Carolina
  - Warner Chilcott Investigational Site, Wilmington, North Carolina
  - Warner Chilcott Investigative Site, Wilmington, North Carolina
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Cincinnati, Ohio
  - Warner Chilcott Investigational Site, Cleveland, Ohio
  - Warner Chilcott Investigational Site, Bala-Cynwyd, Pennsylvania
  - Warner Chilcott Investigational Site, Jenkintown, Pennsylvania
  - Warner Chilcott Investigational Site, Lancaster, Pennsylvania
  - Warner Chilcott Investigational Site, Greer, South Carolina
  - Warner Chilcott Investigational Site, Mt. Pleasant, South Carolina
  - Warner Chilcott Investigational Site, Myrtle Beach, South Carolina
  - Warner Chilcott Investigational Site, Arlington, Texas
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Sugar Land, Texas
  - Warner Chilcott Investigational Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Site, Norfolk, Virginia
  - Warner Chilcott Investigational Site, Richmond, Virginia
  - Warner Chilcott Investigational Site, Mountlake Terrace, Washington
  - Warner Chilcott Investigational Site, Spokane, Washington